CLINICAL TRIAL: NCT01090648
Title: A Study to Survey the Swallowability of Uncoated 200-mg Tablets of Etravirine in HIV-1 Infected Subjects
Brief Title: TMC125HIV1083 - Swallowability of Uncoated 200 mg Etravirine Tablets in HIV-1 Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: CR017038
Record Dates: First submitted 2010-03-11; First posted 2010-03-22 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: HIV-Infections
Keywords: TMC125HIV1083; TMC125; HIV; Etravirine; ETR; Intelence; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — etravirine

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- 001 (Experimental): etravirine One etravirine (ETR) 200 mg uncoated oral tablet and one etravirine (ETR) 200 mg film-coated tablet
  Interventions: Drug: etravirine

INTERVENTIONS:
Drug: etravirine — One etravirine (ETR) 200 mg uncoated oral tablet and one etravirine (ETR) 200 mg film-coated tablet

SUMMARY:
This trial is designed to assess the swallowability of uncoated and film-coated 200 mg etravirine tablets in HIV-1 infected patients. In addition, comparisons between a single 200 mg tablet versus two 100 mg formulations will be made. The outcome of the trial will aid in making decisions about the future commercial 200 mg formulation.

DETAILED DESCRIPTION:
This trial is designed to elicit the swallowability of two formulations of 200 mg tablets of etravirine (ETR). The trial will allow the assessment of the swallowability of the 200 mg uncoated tablet, the 200 mg film-coated tablet and make comparisons between these tablets and with the current commercially available 100 mg (uncoated) tablets. The trial will be performed in HIV-1 infected patients who are currently taking etravirine (ETR) at a total daily dose of 400 mg (four 100 mg tablets, as whole tablets orally) as part of an antiretroviral regimen with virologic suppression (< 50 copies/mL for at least three months). The trial includes only patients who are already taking etravirine since these patients will have pill taking experience and will also have experience with the commercially available 100 mg tablet formulation. A minimum of 45 patients will be included in the trial to assure a sample representative of the HIV-1 infected population. Patients will be given a single dose of the etravirine (ETR) uncoated 200 mg tablet in the morning, and then complete a questionnaire related to that intake. Within 30 minutes, they will be administered the coated 200 mg formulation, followed by a questionnaire. Assessments of the 200 mg tablets will be made in a single-blinded fashion. As the patient will be administered two 200mg tablets in the morning, he/she does not need to take an evening dose on the day of these assessments. The questionnaire will be used to assess swallowability of the 200 mg formulations and of their current 100 mg tablets, and will also evaluate patient preferences. Patients will be followed up for safety and tolerability for one week due to the short duration the patient will be on study treatment; it will be difficult to distinguish between Adverse Events (AEs) resulting from their current etravirine (ETR) intake (four 100 mg tablets) versus the study intake (two 200 mg tablets). A single dose of an etravirine uncoated 200 mg tablet in the morning, followed by completion of a questionnaire related to that intake. Within 30 minutes, patients will be administered the coated 200 mg formulation, again followed by a questionnaire. Maximum 2 weeks screening, 1 day treatment, 1 week follow up. Total duration of participation is 2 weeks maximum.

ELIGIBILITY:
Inclusion Criteria:

* Women must be postmenopausal for at least 2 years, OR be surgically sterile (have had a total hysterectomy or bilateral oophorectomy, tubal ligation/bilateral tubal clips without reversal operation, or otherwise be incapable of becoming pregnant), OR be not heterosexually active for the duration of the study or have a vasectomized partner (confirmed sterile) OR if of childbearing potential and heterosexually active, be practicing a highly effective method of birth control (as specified below) before entry, and agree to continue to use a highly effective method of contraception throughout the study. Women with tubal ligation are required to use one contraceptive method (Note: A male and female condom should not be used together due to risk of breakage or damage caused by latex friction)
* All women must have a negative serum or urine pregnancy test at screening. Women of childbearing potential must have a negative urine pregnancy test at other visits
* Men must agree to use a highly effective method of birth control (i.e., male condom with either female intrauterine device, diaphragm, cervical cap or non-estrogen hormonal based contraceptives) and to not donate sperm during the study
* Patients must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Patient can comply with the protocol requirements

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, would compromise the study or the well-being of the patient or prevent the patient from meeting or performing study requirements
* Any active clinically significant disease (e.g., pancreatitis, cardiac dysfunction) or findings during screening of medical history, laboratory or physical examination that, in the investigator's opinion, would compromise the patient's safety, ability to swallow, or outcome of the trial
* Pregnant or breastfeeding female patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Questionnaire using a 7-point scale to determine the acceptability of swallowing an uncoated 200 mg etravirine (ETR) tablet | Assessment visit (Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- See also: A study to survey the swallowability of non-coated 200-mg tablets of etravirine in HIV-1 infected subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1037&filename=CR017038_CSR.pdf